CLINICAL TRIAL: NCT04657068
Title: A Phase I/IIa, Open-label, Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the ATR Kinase Inhibitor ART0380 Administered Orally as Monotherapy and in Combination to Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of ART0380 for the Treatment of Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Artios Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ART0380C001
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer; Metastatic Cancer; Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Endometrial Cancer; Metastatic Colorectal Cancer; Pancreatic Ductal Adenocarcinoma; Acinar Cell Carcinoma
Keywords: Loss of Ataxia Telangiectasia Mutated (ATM) protein
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms; Carcinoma, Acinar Cell; Hereditary Sensory and Autonomic Neuropathies | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A1 (Experimental): Part A1 evaluated intermittent and continuous dosing of ART0380 monotherapy. Treatment was given in 21-day cycles.
  Interventions: Drug: ART0380
- Part A2 (Experimental): Part A2 evaluated intermittent dosing of ART0380 in combination with gemcitabine in 21-day cycles.
  Interventions: Drug: ART0380; Drug: Gemcitabine
- Part A3 (Experimental): Part A3 evaluated intermittent dosing of ART0380 in combination with irinotecan in 21-day cycles.
  Interventions: Drug: ART0380; Drug: Irinotecan
- Part B1 (Experimental): In Part B1, up to 7 cohorts enrolled participants with solid cancers with alterations in the ATM (ataxia-telangiectasia mutated) gene likely to predict for loss of ATM protein will be treated with either
  * ART0380 monotherapy Or
  * ART0380 in combination with irinotecan
  Interventions: Drug: ART0380; Drug: Irinotecan
- Part B2 (Experimental): In Part B2, participants with high grade serous ovarian, primary peritoneal, or fallopian tube carcinoma were randomized (open label) 1:1 to either ART0380 in combination with gemcitabine or gemcitabine alone.
  Interventions: Drug: ART0380; Drug: Gemcitabine
- Part B3 (Experimental): in Part B3, participants with persistent or recurrent endometrial cancer (EC) received ART0380 monotherapy on either a continuous daily dose or on an intermittent schedule for a 21-day cycle.
  Interventions: Drug: ART0380
- Part B4 (Experimental): In Part B4, participants with advanced or metastatic solid tumors received ART0380 monotherapy on either a continuous daily dose or on an intermittent schedule for a 21-day cycle.
  Interventions: Drug: ART0380
- Part B5 (Experimental): In Part B5, participants with colorectal cancer (CRC) will receive ART0380 in combination with irinotecan on a 21-day cycle.
  Interventions: Drug: ART0380; Drug: Irinotecan
- Part B6 (Experimental): In Part B6, participants with pancreatic ductal adenocarcinoma (PDAC) or acinar cell carcinoma will receive ART0380 in combination with irinotecan on a 21-day cycle.
  Interventions: Drug: ART0380; Drug: Irinotecan
- Part A3 Fed/Fast (Experimental): Part A3 Fed/Fast will evaluate intermittent dosing of ART0380 in combination with irinotecan in 21-day cycles in a fasting or fed state.
  Interventions: Drug: ART0380; Drug: Irinotecan
- Part B7 (Experimental): In Part B7, participants with colorectal cancer (CRC) will receive ART0380 in combination with irinotecan on a 21-day cycle.
  Interventions: Drug: ART0380; Drug: Irinotecan

INTERVENTIONS:
Drug: ART0380 — Participants will receive ART0380 by mouth either intermittently (either once daily 3 days on, 4 days off; days 2-4 and 9-11;or days 1-3 and 8-10) or continuously (once daily each day) in 21 day cycles.
Drug: Gemcitabine — Gemcitabine was administered on Days 1 and 8 of a 21-day cycle.
  Other Names: Gemzar
  Arms: Part A2; Part B2
Drug: Irinotecan — Irinotecan will be administered as a 90-minute infusion on Days 1 and 8 of a 21 day cycle.
  Other Names: Camptosar; Camptothecin-11
  Arms: Part A3; Part A3 Fed/Fast; Part B1; Part B5; Part B6; Part B7

SUMMARY:
This clinical trial is evaluating a drug called ART0380 in participants with advanced or metastatic solid tumors. The main goals of this study are to:

* Find the recommended dose of ART0380 that can be given safely to participants alone and in combination with gemcitabine or irinotecan
* Learn more about the side effects of ART0380 alone and in combination with gemcitabine or irinotecan
* Learn more about the effectiveness of ART0380 alone and in combination with gemcitabine or irinotecan

DETAILED DESCRIPTION:
ART0380 is a new investigational medicinal product that is a potent and selective inhibitor of Ataxia telangiectasia and Rad3-related (ATR). ART0380 is being developed as an oral anti-cancer agent for the treatment of participants with cancers that harbor defects in deoxyribonucleic acid (DNA) repair and in combination with agents including those that cause DNA damage.

This study is an open-label Phase I/IIa study designed to evaluate the safety, tolerability, PK and preliminary efficacy of ART0380 as monotherapy or in combination with gemcitabine or irinotecan in participants with advanced or metastatic solid tumors, advanced or solid tumors that fail to express Ataxia-Telangiectasia Mutated protein kinase (ATM) by immunohistochemistry, and high grade serous ovarian, primary peritoneal or fallopian tube carcinoma.

ELIGIBILITY:
General Inclusion Criteria:

* Signed informed consent
* Discontinued all previous treatments for cancer for at least 21 days or 5 half-lives, whichever is shorter, and recovered from the acute effects of therapy to CTCAE Grade ≤1. Palliative radiotherapy must have completed 1 week prior to start of study treatment.
* If patients have a known germline BRCA mutation or a cancer with a somatic BRCA mutations or which is HRD positive and for which there is an approved PARP inhibitor, participants should have received such treatment before participating in the study unless contra-indicated
* At least 1 radiologically evaluable lesion (measurable and/or non-measurable) that can be assessed at baseline and is suitable for repeated radiological evaluation by RECIST v1.1 or Prostate Cancer Working Group-3 Guidelines (PCWG-3)
* Acceptable hematologic, renal, hepatic, and coagulation functions independent of transfusions and granulocyte colony-stimulating factor
* Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis.
* Female patients of childbearing potential and male patients with female partners of childbearing potential are required to use highly effective contraception plus one barrier method during their participation in the study and for 7 months and 5 months respectively following the last dose. For male and female patients given gemcitabine or irinotecan, highly effective contraception plus one barrier method must be used from study entry until 6 months after the last dose of study treatment. Male patients are required to refrain from donating sperm and female patients are required to refrain from donating eggs, during their participation in the study and for 6 months following last dose.
* Estimated life expectancy of ≥12 weeks
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Performance status of 0-1 on the ECOG Scale

Additional inclusion criteria for participants in dose escalation (Part A1):

* Advanced or metastatic cancer which is refractory to standard therapies, or for which no standard therapies exist, or for which the investigator feels no other active therapy is required for the duration of the study
* Performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale

Additional inclusion criteria for participants in dose escalation (Part A2):

•Advanced or metastatic cancer for which gemcitabine is an appropriate treatment. Prior treatment with gemcitabine is permitted.

Additional inclusion criteria for participants in dose escalation (Part A3):

* Advanced or metastatic cancer for which irinotecan is an appropriate treatment. Prior treatment with irinotecan is permitted.
* For food effect cohort only: Patients must be able to eat a high-fat meal within a 30 minute period, as provided by the study site.

Additional inclusion criteria for participants in dose expansion (Part B1):

* Patients with advanced or metastatic solid tumors with alterations to the ATM gene likely to predict for loss of ATM protein
* Have at least 1 measurable lesion assessable using standard techniques by RECIST v1.1
* For France only ART0380 Monotherapy; Patient that is not eligible for curative treatment, for whom all standard of care therapies have failed and no therapies known to provide clinical benefit are available.
* Combination arms; Patients for which irinotecan is an appropriate treatment. Prior treatment with irinotecan is permitted.
* For Spain only ART0380 Combination therapy, Patient that is not eligible for curative treatment, for whom standard of care therapies have failed.

Additional inclusion criteria for participants in dose expansion (Part B2):

* Patients with a known germline BRCA mutation, or a cancer with a known somatic BRCA mutation, or which is known to be HRD positive, and for which there is an approved PARP inhibitor should have received such treatment before participating in the study, unless contra-indicated.
* Females with histologically-confirmed diagnosis of high grade serous carcinoma of the ovary, fallopian tube or primary peritoneum that is not amenable to curative therapy
* Platinum-resistant disease, defined as disease progression within 6 months of last receipt of platinum-based chemotherapy. Patients must not have had primary platinum-refractory disease (disease that progressed during first-line platinum-based therapy).
* No more than one prior regimen in the platinum-resistant setting. Hormonal therapies and antiangiogenic therapies (as single agents) and PARP inhibitors used as maintenance therapy are not considered as separate lines of therapy. Patients should have previously received bevacizumab and chemotherapy unless contra-indicated.
* Have not received prior treatment with gemcitabine unless administered in combination with a platinum with no disease progression within 12 months after completion of that regimen
* Have at least 1 measurable lesion assessable using standard techniques by RECIST v1.1

Inclusion criteria specific to Part B3

* Persistent or recurrent endometrial cancer with biological selection.:
* Patients should have received taxane/platinum chemotherapy, unless contraindicated.
* Measurable disease.

Inclusion criteria specific to Part B4

* Advanced or metastatic solid cancers of any histology with biological selection
* If a PD-1/PDL-1 inhibitor (eg, pembrolizumab) is approved and available for the patient's cancer, the patient should have received such treatment before participating in this study.
* Radiologically evaluable disease
* Performance status of 0-1 on the ECOG scale

Inclusion criteria specific to Part B5 and B7

* Metastatic CRC with alterations to the ATM gene
* Participants should have previously received appropriate prior lines of therapy in this setting.
* Have at least 1 measurable lesion assessable using standard techniques by RECIST v1.1.
* Part B5 (3L) only:
* Patients must have received a maximum of exactly 2 prior chemotherapy regimens for the treatment of CRC which must have included a fluoropyrimidine, oxaliplatin and irinotecan unless contraindicated or unavailable
* Part B7 (2L) only:
* Patients must have received exactly 1 prior chemotherapy regimen for the treatment of CRC which must have included a fluoropyrimidine unless contraindicated or unavailable

Inclusion criteria specific to Part B6:

* Metastatic or locally advanced PDAC or acinar cell carcinoma with alterations to the ATM gene
* Participants should have previously received prior lines of therapy in this setting
* Have at least 1 measurable lesion assessable using standard techniques by RECIST v1.1
* Serum albumin ≥3g/dL within 7 days prior to first dose.

General Exclusion Criteria:

* Women who are pregnant, breast feeding, or who plan to become pregnant while in the study or within 7 months after the last administration of study treatment
* Men who plan to father a child while in the study or within5 months after the last administration of study treatment
* Serious concomitant systemic disorder that would compromise the participants ability to adhere to the protocol including: one or more opportunistic HIV/AIDs-related infections within the past 12 months, a known hepatitis B virus, or known hepatitis C virus; documented active or chronic tuberculosis infection; malignancy prior to the one currently being treated that is not in remission
* Have ongoing interstitial lung disease or pneumonitis (whether symptomatic or asymptomatic).
* Moderate or severe cardiovascular disease
* Valvulopathy that is severe, moderate, or deemed clinically significant
* Documented major electrocardiogram (ECG) abnormalities which are clinically significant
* Symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment
* Received a live vaccine within 30 days before the first dose of study treatment
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate
* Recent major surgery within 4 weeks prior to entry into the study or minor surgery within 1 week of entry into the study
* Significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 12 weeks prior to enrollment
* Currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study

Additional exclusion criteria for participants in dose escalation (Part A3, B1, B5, B6, and B7 in combination with irinotecan):

* Patients who have symptoms or signs of clinically unacceptable deterioration of the primary disease at the time of screening.
* Patients receiving inhibitors of UGT1A1 within 2 weeks before the first dose of study treatment
* Part A3 Fed-fasted cohort only: Patients receiving acid reducing agents within 1 week before the first dose of study treatment will be excluded
* Part B6 only: Neuroendocrine (carcinoid, islet cell) or adenosquamous carcinoma pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2020-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Maximum tolerated dose (MTD) by the number of participants with dose limiting toxicities (DLTs) from ART0380 monotherapy and in combination with gemcitabine or irinotecan | From Cycle 0 Day -2 to Cycle 1 Day 21. Each cycle is 21 days.
Parts B1/B3/B4: Number of participants with adverse events following administration of ART0380 monotherapy and/or in combination with irinotecan at RP2Ds. | From Cycle 1 Day 1 until up to 30 days after the last dose of ART0380. Each cycle is 21 days.
  Safety reported as incidence of adverse events
Part B2: Progression free survival by RECIST 1.1 in participants receiving ART0380 in combination with gemcitabine or gemcitabine alone | Every 6 weeks from Cycle 1 Day 1 for 18 weeks, then every 9 weeks up to approximately 24 months. Each cycle is 21 days.
  Progression free survival (PFS)
Parts B5/B6/B7: Object Response Rate (ORR) based on RECIST 1.1 to access anti-tumor activity of ART0380 in combination with irinotecan in each cohort. | Every 6 weeks from Cycle 1 Day 1, until disease progression or death or start of a new anti-cancer therapy, up to 2 years. Each Cycle is 21 days.
  Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Part B2: Number of participants with adverse events following administration of ART0380 in combination with gemcitabine or gemcitabine alone | From Cycle 1 Day 1 until up to 30 days after the last dose of ART0380 or gemcitabine. Each cycle is 21 days.
Part B5/B6/B7: Number of participants with adverse events following administration of ART0380 at the RP2D in combination with irinotecan. | From Cycle 1 Day 1 until up to 30 days after the last dose of ART0380 or irinotecan. Each cycle is 21 days.
Pharmacokinetic Analysis (single dose): determine the plasma concentration of ART0380 when given alone and in combination | PK will be measured at each cycle from Cycle 0 to Cycle 4. Each cycle is 21 days.
Pharmacokinetic Analysis (multiple dose): determine the plasma concentration of ART0380 when given alone and in combination | PK will be measured at each cycle from Cycle 0 to Cycle 4. Each cycle is 21 days.
Pharmacokinetic Analysis: Renal clearance of ART0380 | Urine PK will be measured during Cycle 1. Cycle 1 is 21 days.
Parts A1, A2, A3, B1, B3, B4: Objective response rate based on RECIST 1.1 | Every 6 weeks from Cycle 1 Day 1 for 18 weeks, then every 9 weeks up to approximately 24 months. Each cycle is 21 days.
Parts A1, A2, A3, B1, B3, B4, B5, B6, and B7: Duration of response based on RECIST 1.1 | Every 6 weeks from Cycle 1 Day 1 for 18 weeks, then every 9 weeks up to approximately 24 months. Each cycle is 21 days.
Parts A1, A2, A3, B1, B3, B4, B5, B6, and B7: Progression free survival based on RECIST 1.1 | Every 6 weeks from Cycle 1 Day 1 for 18 weeks, then every 9 weeks up to approximately 24 months. Each cycle is 21 days.
Pharmacokinetic Analysis: Area Under The Curve Plasma Concentration Time Curve from zero to 12 hours (AUC0-12) | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Maximum plasma Concentration (Cmax) in a fasting and fed state. | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Time to Maximum plasma concentration (Tmax) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Area Under The Curve Plasma Concentration Time Curve from zero to the time of last plasma concentration (AUC0-t) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Terminal half-life (t1/2) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Area under the concentration-time curve over the dosing interval (AUC(0-tau)) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Area Under The Curve Plasma Concentration Time Curve over the last 12-h dosing interval (AUC012) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Area under the concentration-time curve over the dosing interval (AUC(0-infinity)) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Area under the concentration-time curve for Oral Clearance (CL/F) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Pharmacokinetic Analysis: Area under the concentration-time curve for Volume of Distribution (Vz/F) in a fasting and fed state | PK will be measured during Cycle 1. Cycle 1 is 21 days
Parts B1/B3/B4/B5/B6/B7: Response and disease progression by Serological tumor markers (CA-19-9, CAE, CA-125, and Prostate Specific Antigen (PSA)). | Tumor markers will be measured for 18 weeks, then every 9 weeks thereafter.
Parts B1/B3/B4/B5/B6/B7: Overall Survival | After first dose through PFS/OS follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, MD, Study Chair — Tennessee Oncology; Antonio Gonzalez, MD, PHD, Study Chair — Clinica Universidad de Navarra, Madrid; Susanna Ulahannan, MD, Principal Investigator — Oklahoma University; Kim Reiss Binder, MD, Principal Investigator — University of Pennsylvania / Abramson Cancer Center
Locations (75):
- United States (40):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic (Arizona), Scottsdale, Arizona
  - University of Arkansas - Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sansum Clinic, Santa Barbara, California
  - Providence Medical Foundation, Santa Rosa, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mayo Clinic (Florida), Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Our Lady of the Lake, Baton Rouge, Louisiana
  - Maryland Oncology Hematology - Primary, Columbia, Maryland
  - Minnesota Oncology Hematology, Maple Grove, Minnesota
  - Mayo Clinic (Minnesota), Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Northwell Health Cancer Institute, Lake Success, New York
  - Oncology Hematology Care Primary, Cincinnati, Ohio
  - Taylor Cancer Research Center, Maumee, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania / Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Clinical Research Organization, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Northeast Texas, Flower Mound, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
- France (2):
  - Institut Gustave Roussy, Villejuif, Cedex
  - Institut Bergonie, Bordeau
- Spain (29):
  - Hospital General Universitario de Elche, Elche, Alicante
  - H. Parc Tauli, Sabadell, Barcelona
  - Next Oncology Barcelona, IOB, Barcelona, Catalonia
  - Hospital Arnau de Vilanova, Lleida, Catalonia
  - Hospital Universitario La Paz, Madrid, Madrid
  - Next - Hospital Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Clínica Universidad de Navarra, Madrid, Planta -2
  - START Rioja, Rioja, Spain
  - Instituto Valenciano de Oncología (IVO), Valencia, Spain
  - Hospital Teresa Herrera (CHUAC), A Coruña
  - Institut Català d'Oncologia Badalona - Hospital Germans Trias i Pujol, Badalona
  - Vall d'Hebron Institute of Oncology (VIHO), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO Hospitalet, Barcelona
  - Hospital Universitario Reina Sofia de Córdoba, Córdoba
  - Hospital Universitari Doctor Josep Trueta- ICO de Girona, Girona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Center (Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - START Madrid Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid (Hospital San Chinarro), Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario De Navarra, Pamplona
  - Hospital Virgen Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Incliva Biomedical Research Institute, University of Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (4):
  - Guy's and St Thomas' NHS Foundation Trust, London, London
  - The Christie NHS Foundation Trust - The Christie Clinic, Manchester, United Kingdom
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Sarah Cannon Research Institute UK, London

IPD SHARING:
Plan to Share IPD: No